CLINICAL TRIAL: NCT06601608
Title: Efficacy of Locally Delivered Rosemary Extract Gel As an Adjunct to Non-Surgical Periodontal Therapy in Management of Periodontitis (A Randomized Controlled Clinical Trial with Microbiological Analysis)
Brief Title: Efficacy of Locally Delivered Rosemary Extract Gel in Management of Periodontitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Roba abdelhamid mohamed elhady, Resident dentist at department of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec IM122331
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Periodontitis (stage 3); Periodontal Pocket
Keywords: Periodontitis; local delivery drug; microbiological analysis
MeSH Terms: conditions — Periodontitis; Periodontal Pocket | interventions — Phytotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rosemary extract gel (Experimental): rosemary extract gel will be applied in deep periodontal pockets with a concentration 5%.
  Interventions: Drug: Herbal therapy
- placebo gel (Placebo Comparator): a placebo gel will be applied in deep periodontal pockets in stage III periodontitis patients as an adjunct to non-surgical periodontal therapy.
  Interventions: Drug: Placebo Drug

INTERVENTIONS:
Drug: Herbal therapy — rosemary extract gel is used for the first time as a local drug delivery as an adjunct to non-surgical periodontal therapy in management of stage III periodontitis patients.
  Other Names: rosemary extract gel; local delivery drug; phytotherapy
  Arms: Rosemary extract gel
Drug: Placebo Drug — a placebo gel will be applied in deep pockets (>5mm) in stage III periodontitis patients as an adjunct to non-surgical periodontal therapy
  Arms: placebo gel

SUMMARY:
Rosemary extract is known for its antibacterial, anti-inflammatory and anti-oxidant properties that make it a promising therapeutic aid as a local delivery drug in deep periodontal pockets in adjunct to non-surgical periodontal therapy in management of periodontitis. These properties are due to the high content of phenolic compounds such as carnosic acid, urolic acid, rosmarinic acid or chlorogenic acid. Rosemary extract was previously investigated and proved its effectiveness against periodontopathogens in-vitro. Thus, its selected for this study to be administered in a gel form to assess its efficacy in management of periodontitis.

DETAILED DESCRIPTION:
Sixteen patients with deep periodontal pockets more than 5 mm will be randomly assigned into 2 equal groups. The test group will receive the rosemary extract gel in adjunct to non-surgical periodontal therapy, while the control group will receive placebo gel.

Clinical evaluation of the clinical parameters including probing depth, gingival index, plaque index and clinical attachment level will be recorded.

Microbiological analysis using PCR test will be performed using perio-papers.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders aged between 25-45 years.
2. Healthy adult patients as evidenced by Burket's oral medicine health history questionnaire.
3. Stage III grade B periodontitis with at least two non-adjacent sites in posterior teeth with PD ≥ 6 mm, CAL ≥ 5 mm showing BOP and ≤ 4 teeth lost due to periodontitis.
4. Patients ready to comply with oral hygiene measures.

Exclusion Criteria:

1. Smokers.
2. Pregnant or lactating females.
3. Drug abusers.
4. Patients taking antibiotics or performed any periodontal treatment in the previous 6 months.
5. Patients who have a known allergy or hypersensitivity to rosemary, its constituents, or other members of the Lamiaceae family.
6. Patients with parafunctional habits.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
probing depth | change from baseline at 3 months
  Will be measured from the gingival margin to the bottom of the periodontal pocket to the nearest mm. with use of UNC 15 periodontal probe.

SECONDARY OUTCOMES:
clinical attachment level, plaque index and gingival index | change from baseline at 3 months
  - Clinical attachment level (CAL): Will be measured from the CEJ to the depth of the periodontal pocket in millimeters.
  * Plaque index:
    0 = No plaque in gingival area.
    1. = A film of plaque adhering to the free gingival margin and adjacent area of tooth.
       The plaque may be recognized only by running a probe across the tooth surface.
    2. = Moderate accumulation of soft deposit within the gingival pocket and on the gingival pocket and on the gingival margin and/or adjacent tooth surface that can be seen by naked eye.
    3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
  * Gingival index:
    0 = Normal gingiva
    1. = Mild inflammation - slight edema. No bleeding on probing
    2. = Moderate inflammation -redness, edema and glazing. Bleeding on probing.
    3. = Severe inflammation - marked redness and edema. Ulceration. Tendency to spontaneous bleeding
microbiological analysis | The bacterial load in the GCF sample will be assessed at baseline, 1 week and 1 month post-operatively.
  Microbiological analysis to evaluate the antibacterial effect of rosemary extract gel on quantitative change of P.gingivalis and A.actinomycetemcomitans in the gingival crevicular fluid (GCF) using perio-papers.
  Analyzed samples will be done using real time PCR technique.

CONTACTS AND LOCATIONS:
Overall Officials: Nevine Hassan Kheir El Din, Professor, Study Director — Faculty of Dentistry - Ain Shams University
Locations (1):
- Faculty of Dentistry - Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided